CLINICAL TRIAL: NCT06878742
Title: Dose-finding for Dobutamine During Transitional Circulation in the Very Preterm Infant
Brief Title: Dose-finding for Dobutamine During Transitional Circulation in Very Preterm Infants
Acronym: NeoCirc-002
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP 6422
Record Dates: First submitted 2024-12-02; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Infant, Premature, Diseases; Circulatory and Respiratory Physiological Phenomena
Keywords: Hemodynamic insuffiency; Low superior vena cava flow
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Intervention Model Description: NeoCirc-002 is a single center, dose finding trial to define the minimum effective dose of dobutamine to treat early hemodynamic insufficiency in the preterm infant (less than 33 completed weeks' gestation), defined as presence of low SVC flow (<51 ml/k/min) within the first 72 hours from birth.
  The trial is a low-intervention clinical trial since dobutamine is the standard treatment for circulatory failure in preterm infants during transitional circulation, the dosages studied are within the standard therapeutic range, and the diagnostic supplementary procedures are in routine clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dobutamine dose A (Experimental): Intravenous dobutamine will be administered at a dose of 5 mcg/kg/min. Weaning and stopping of the dobutamine infusion will be determined by the attending physician, following local policies.
  Interventions: Drug: Intravenous dobutamine 5 mcg/kg/min
- Dobutamine dose B (Experimental): Intravenous dobutamine will be administered at a dose of 7.5 mcg/kg/min. Weaning and stopping of the dobutamine infusion will be determined by the attending physician, following local policies.
  Interventions: Drug: Intravenous dobutamine 7.5 mcg/kg/min
- Dobutamine dose C (Experimental): Intravenous dobutamine will be administered at a dose of 10 mcg/kg/min. Weaning and stopping of the dobutamine infusion will be determined by the attending physician, following local policies.
  Interventions: Drug: Intravenous dobutamine 10 mcg/kg/min
- Dobutamine dose D (Experimental): Intravenous dobutamine will be administered at a dose of 12.5 mcg/kg/min. Weaning and stopping of the dobutamine infusion will be determined by the attending physician, following local policies.
  Interventions: Drug: Intravenous dobutamine 12.5 mcg/kg/min
- Dobutamine dose E (Experimental): Intravenous dobutamine will be administered at a dose of 15 mcg/kg/min. Weaning and stopping of the dobutamine infusion will be determined by the attending physician, following local policies.
  Interventions: Drug: Intravenous dobutamine 15 mcg/kg/min

INTERVENTIONS:
Drug: Intravenous dobutamine 5 mcg/kg/min — Intravenous dobutamine will be administered at a dose of 5 mcg/kg/min.
  Arms: Dobutamine dose A
Drug: Intravenous dobutamine 7.5 mcg/kg/min — Intravenous dobutamine will be administered at a dose of 7.5 mcg/kg/min.
  Arms: Dobutamine dose B
Drug: Intravenous dobutamine 10 mcg/kg/min — Intravenous dobutamine will be administered at a dose of 10 mcg/kg/min.
  Arms: Dobutamine dose C
Drug: Intravenous dobutamine 12.5 mcg/kg/min — Intravenous dobutamine will be administered at a dose of 12.5 mcg/kg/min.
  Arms: Dobutamine dose D
Drug: Intravenous dobutamine 15 mcg/kg/min — Intravenous dobutamine will be administered at a dose of 15 mcg/kg/min.
  Arms: Dobutamine dose E

SUMMARY:
Single centre, dose finding trial to establish the minimum effective dose of dobutamine required to treat hemodynamic insufficiency, defined as low superior vena cava (SVC) flow, in infants below 33 weeks' gestation during transitional circulation (first 72 hours from birth).

ELIGIBILITY:
Inclusion Criteria:

* Born with up to 32(+6) weeks gestation
* Presence of hemodynamic insufficiency, defined as SVC flow <51 ml/kg/min.
* Provision of signed and dated informed consent form by father/mother or legally designated representative, which can be given antenatally.

Exclusion Criteria:

* Neonates considered non-viable, with a clinical decision not to provide life support
* Infants with severe congenital hydrops fetalis needing chest or peritoneal drainage before recruitment
* Infants already on dobutamine treatment
* Infants with congenital malformations likely to affect cardiovascular adaptation (including: congenital diaphragmatic hernia, gastroschisis or congenital heart defects)
* Infants with chromosomal anomalies
* Lack of parental signed informed consent

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Minimum dobutamine dose to reach and maintain a SVC flow above 55 ml/kg/min | 1 and 3 hours
  Short-term pharmacodynamics (PD) endpoint: Minimum dobutamine dose to reach and maintain a superior vena cava (SVC) flow above 55 ml/kg/min on an echocardiogram performed at 1 and 3 hours after effective infusion of the allocated dose.
  The effective start of the infusion (t0) will be calculated as the time at which the infusion pump is switched on plus the empirical value for the interval arising from the dead space. We summarize t0 as "the time at which dobutamine is expected to reach the circulation"

SECONDARY OUTCOMES:
Proportion of neonates achieving and maintaining a clinically acceptable haemodynamic status | 72 hours
  Proportion of neonates achieving and maintaining a clinically acceptable haemodynamic status with the dobutamine infusion alone in the first 72 hours from birth.
  Acceptable hemodynamic status is defined as the achievement and maintenance of dose success during the first 72 h from birth. The loss of such acceptable haemodynamic status occurs whenever there is a change in therapeutic strategy that involves cardiovascular treatment other than dobutamine alone due to exceeded safety parameters, treatment failure of the investigational infusion or the need for rescue treatment or death; any additional fluid bolus is considered as cardiovascular treatment.
Absolute and relative frequencies of adverse events and severe adverse events | Through study completion, an average of 12 months
  Absolute and relative frequencies of adverse events (AEs) and severe adverse events (SAEs), to be recorded and compared between groups.
  AEs are defined as any untoward medical occurrence in a patient or clinical investigation patients administered a medicinal product, which does not necessarily have a causal relationship with this treatment (the study medication).
  SAEs are defined as any untoward medical occurrence that at any dose:
  * Results in death,
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital anomaly/birth defect.
  * Other important medical events.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario Quironsalud, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No